CLINICAL TRIAL: NCT06696417
Title: A Prospective, Single-arm, Multicenter, Phase IV Study to Evaluate the Efficacy and Safety of Vunakizumab in Adults With Moderate-to-severe Plaque Psoriasis Who Have Not Previously Received Biologics
Brief Title: Phase IV Study: Vunakizumab Efficacy and Safety in Moderate-to-severe Plaque Psoriasis
Status: Recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Gao Xinghua, Distinguished Professor of Cheung Kong Scholars；Vice President, First Affiliated Hospital of China Medical University, First Hospital of China Medical University
Other Study IDs: MA-DER-RWS-001
Record Dates: First submitted 2024-11-12; First posted 2024-11-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Weeks
Biospecimen Retention: Samples Without DNA — This study only collects routine testing data and does not specifically collect biospecimens.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Drug group：vunakizumab (IL-17A inhibitor) — The recommended dose of vunakizumab was 240 mg, administered subcutaneously at weeks 0, 2, and 4, then every 4 weeks, with a final injection at 48 weeks

SUMMARY:
This is a multicenter, prospective, observational study of 1516 patients with moderate-to-severe chronic plaque psoriasis to evaluate the efficacy and safety of vunakizumab in patients with moderate-to-severe chronic plaque psoriasis. Approximately 50-100 clinical trial centers are planned to participate in the study. The study consisted of a 7-day screening period, a 52-week treatment period and an 8-week safety follow-up period.

The recommended dose of vunakizumab is 240 mg (120 mg in two injections), with subcutaneous injection at week 0, 2, and 4, followed by a dose every 4 weeks and a final injection at week 48 (the actual treatment regimen is based on the clinician's recommendation). After the corresponding assessment at 52 weeks, an 8-week safety follow-up period was entered until the end of the study.

DETAILED DESCRIPTION:
The vunakizumab is a humanized IL-17A inhibitor with innovative binding epitopes, which accurately binds to IL-17A, the core pathogenic factor of psoriasis. However, there is still a lack of efficacy and safety data in a large sample size of the Chinese population after marketing. Therefore, this study is intended to observe the efficacy and safety of vunachizumab in a larger population. The clinical efficacy of vunakizumab on special sites and the influence of comorbidity on the treatment of psoriasis are also paid attention to. At the same time, the improvement effect of vunakizumab on the quality of life and mental health of psoriasis patients is explored through patient-reported outcome (PRO) and patient satisfaction survey, so as to develop a clinical program that can benefit psoriasis patients physically and mentally.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old at the time of signing the informed consent, regardless of gender;
* Moderate to severe plaque psoriasis was diagnosed;
* Plan to receive vunakizumab therapy as assessed by the investigator;
* The subject voluntarily signs informed consent before the start of any procedures related to the study, can communicate with the researcher smoothly, understands and is willing to strictly comply with the requirements of this clinical study protocol to complete the study; Patients voluntarily sign informed consent forms.

Exclusion Criteria:

* Previous treatment with biological agents: including but not limited to anti-tumor necrosis factor-α (TNF-α), anti-IL-17, anti-IL-17 receptor, anti-IL-12 /IL-23 or IL-23p19 antibody drugs;
* Severe hypersensitivity to vunakizumab active ingredient or any excipients;
* Patients with clinically important active diseases, such as active tuberculosis, active hepatitis, and active malignant tumors;
* Fertile women (defined as all women with physical conditions necessary for pregnancy) and men who are pregnant or unwilling or unable to use highly effective birth control during the study period and within 20 weeks after last receiving the study drug;
* Any other circumstances that the investigator believes will prevent the subject from following and completing the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate and severe plaque psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 1516 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
The overall clinical clearance rate of skin lesions | Three months
  1. The proportion of subjects who achieved at least a 90% improvement from baseline in PASI scores by week 12 (PASI 90). (PASI: Psoriasis Area and Severity Index, 0 ≤ PASI ≤ 72, where a higher score indicates a greater extent of the disease and more severe skin lesion severity.)
  2. Proportion of subjects achieving sPGA 0/1 response at week 12. (sPGA 0/1 response is defined as an sPGA score of 0 (clear) or 1 (almost clear))

SECONDARY OUTCOMES:
The overall clinical clearance rate of skin lesions | One month， Three months，Twelve months
  Proportion of subjects with PASI 75, PASI 90, PASI 100, sPGA 0/1, and sPGA 0 at week 4, 12, and 52.
The time when subjects reached PASI 75 and PASI 90 within 12 weeks | Three months
The time when subjects reached PASI 75, PASI 90, PASI 100 at 52 weeks. | Twelve months
Changes in PASI scores relative to baseline at each visit point during 52 weeks. | Twelve months
Response rates of ACR (American College of Rheumatology) 20, ACR50 and ACR70 at week 4, 12, 24 and 52. | One month， Three months， Six months，Twelve months
  ACR20 refers to the improvement of at least 20% in the number of swollen and tender joints in rheumatoid arthritis treatment, along with improvement of at least 20% in at least three of the other five assessment criteria. ACR50 and ACR70 are defined using the same criteria, representing a 50% and 70% improvement, respectively.
Weeks 12 and 52 Treatment Satisfaction Questionnaire for Medication (TSQM) survey questionnaire. | Three months，Twelve months
  0 ≤ TSQM ≤ 100, where a higher score indicates greater patient satisfaction with the medication

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China